CLINICAL TRIAL: NCT05322278
Title: Obstetric Outcomes After Double Embryo Transfer in Intracytoplasmic Sperm Injection
Brief Title: Obstetric Outcomes After Double Embryo Transfer
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Shehata Mohamed Ismail, Faculty of medicine, Assiut University, 71515 Assiut, Egypt, Assiut University
Other Study IDs: DET in ICSI
Record Dates: First submitted 2021-12-12; First posted 2022-04-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Double-Embryo Transfer in ICSI
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Single Embryo Transfer: Single Embryo Transfer
  Interventions: Other: Data collection
- Double embryo transfer
  Interventions: Other: Data collection
- 3 embryo transfer
  Interventions: Other: Data collection
- 4 embryo transfer
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — No interventions

SUMMARY:
Aim ; to compare obstetric outcomes in relation to number of embryo transfer in ICSI

DETAILED DESCRIPTION:
Assisted reproductive technology with intracytoplasmic sperm injection (ICSI) and IVF is becoming an international direction for couples struggling with infertility. The increasing popularity and frequency of these techniques and the data generated from it has given us a better overview of the efficacy, consequences and costs of these techniques.

The aim of assisted reproductive technology (ART) is to achieve pregnancy while decreasing the risk of multiple gestations. When compared with elective single embryo transfer (SET), double embryo transfer (DET) demonstrates a superior pregnancy and live birth rate with a significantly higher risk of multiple gestations. The high frequency of multiple births is the main factor which leads to adverse outcome in IVF/intracytoplasmic sperm injection (ICSI) treatment. Transfer of two embryos does not diminish the chance of a birth when compared with three embryo transfer. How would be the obstetric outcome in pregnancies resulting from DET in IVF/ICSI cycles.

Despite achieving a higher pregnancy rates, DET in ART leads to an increase in multiple gestation pregnancies, which are associated with increased both maternal and neonatal morbidity and mortality.

Twin pregnancies have a higher incidence of preterm cesarean sections , admissions to the neonatal intensive care unit (NICU), and other maternal complications, when compared with singleton pregnancies. Twin pregnancies have a higher incidence of preterm cesarean sections , admissions to the neonatal intensive care unit (NICU), and other maternal complications, when compared with singleton pregnancies.

Most patients prefer to have two embryos transferred, due to financial considerations being the main reason.

Studies demonstrate that patients are more likely prefer to choose SET when educated about the risks of multiple gestation pregnancy, but select two embryos for transfer if they have a lower pregnancy rate when compared with transferring one embryo .

Cost effectiveness research comparing single versus DET after in vitro fertilization (IVF) has previously been performed, with most studies taking place in areas with mandated IVF insurance coverage, and few incorporating hospital costs linked to obstetrical and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* all patients subjected with ICSI pregnancy

Exclusion Criteria:

* incomplete data

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All women have ICSI at IVF unit at AUH
Sampling Method: Non-Probability Sample
Enrollment: 927 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Live birth | 1 year
  Comparison

SECONDARY OUTCOMES:
Rate of miscarriage | 1 year
  Comparison
Rate of neonatal morbidities and mortalities in single embryo transfer versus double embryo transfer | 1 year
  Comparison
Rate of admission to NICU | 1 year
  Comparison
Rate of multiple pregnancies | 1 year
  Comparison
Rate of preterm | 1 year
  Comparison
Rate of PPROM | 1 year
  Comparison
Rate of Clinical pregnancy | 1 year
  Comparison
Rate of chemical pregnancy | 1 year
  Comparison

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Mohamed Abd Elmageed Badran, Lecturer, Study Chair — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clua E, Roca-Feliu M, Tresanchez M, Latre L, Rodriguez I, Martinez F, Barri PN, Veiga A. Single or double embryo transfer? Decision-making process in patients participating in an oocyte donation program. Gynecol Endocrinol. 2020 Apr;36(4):365-369. doi: 10.1080/09513590.2019.1653845. Epub 2019 Aug 29. PMID 31464145
- [Background] Gremeau AS, Brugnon F, Bouraoui Z, Peikhrishvili R, Janny L, Pouly JL. [Outcome of elective single or double embryo transfer in first and second IVF/ICSI cycles]. Gynecol Obstet Fertil. 2011 Feb;39(2):70-5. doi: 10.1016/j.gyobfe.2010.08.005. French. PMID 21316284